CLINICAL TRIAL: NCT05988840
Title: Acquisition and Analysis of Relationships Between Longitudinal Emotional Signals Produced by an Artificial Intelligence Algorithm and Self-questionnaires Used in the Psychiatric Follow-up of Patients With Mood and/or Anxiety Disorders: a Real-Environment Study.
Acronym: EMOACQ-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Emobot (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A01589-36
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Anxiety Disorders; Major Depressive Disorder
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The hardware group (on-board camera): A physical device equipped with a camera and embedding the acquisition/monitoring software. Positioned in the living space, it will be possible to capture the facial expressions of the person in ecology, for example when watching a TV program or reading.
  Interventions: Other: Acquisition and analysis of relationships between Longitudinal Emotional Signals produced by a software and Self-questionnaires.
- The software-only group (running on a PC or tablet and using the available webcam): Software running on a computer, connected to the computer's camera (webcam). If the person is teleworking on a PC, it is expected that images will be captured during videoconferencing-type interactions.
  Interventions: Other: Acquisition and analysis of relationships between Longitudinal Emotional Signals produced by a software and Self-questionnaires.

INTERVENTIONS:
Other: Acquisition and analysis of relationships between Longitudinal Emotional Signals produced by a software and Self-questionnaires. — Using the tool developed by Emobot, EMOACQ-1 is a study that passively and non-interventionaly collects data by capturing patients' facial expressions throughout the day, and then measures the correlation between emotional signals and the results of measurement questionnaires used in psychiatry.

SUMMARY:
The worldwide prevalence of anxiety and depression increased massively during the pandemic, with a 25% rise in the number of patients suffering from psychological distress. Psychiatrists, and even more so general practitioners, need measurement tools that enable them to remotely monitor their patients' psychological state of health, and to be automatically alerted in the event of a break in behavior.

In this study, the investigators propose to collect clinical data along with longitudinal measurement of patients' emotions. Emobot proposes to analyze the evolution of mood disorders over time by passively studying people's emotional behavior. The aim of EMOACQ-1 is to acquire knowledge and produce a quantitative link between emotional expression and mood disorders, ultimately facilitating the understanding and management of these disorders.

Through this study, could be developed a technological solution to support healthcare professionals and patients in psychiatry, a field known as the "poor relation of medicine" and lacking in resources. Such a solution would enable better understanding, disorders remote & continuous monitoring and, ultimately, better treatment of these disorders.

The investigators will process the data by carrying out a number of analyses, including descriptive, comparative and correlation studies of the data from the self-questionnaire results and the emotional signals captured by the devices.

Finally, the aim will be to predict questionnaire scores from the emotional signals produced.

ELIGIBILITY:
Inclusion Criteria:

* Persons over the age of 18 who volunteer to take part in research
* Must have access to a computer with an Internet connection,
* Written comprehension of French.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The first cohort of 20 participants will be provided with the 20 measuring embedded device, we will be able to collect specific data at targeted times and for specific activities.
  The second cohort formed with the remaining participants will receive the software on their personal computer, enabling us to capture more general data and analyze behavior patterns in less controlled contexts.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-17 (Estimated); Primary Completion 2024-08-17 (Estimated); Study Completion 2024-10-17 (Estimated)

PRIMARY OUTCOMES:
Repeated measurements Correlations between emotional signals and studied disorders standardized tests. | 10 months
  Repeated measurements Correlations between emotional signals and studied disorders standardized tests.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: D. Agarwal et al. From Multimodal to Unimodal Attention in Transformers using Knowledge Distillation. Nov 2021, Virtual, United States. — https://hal.science/hal-03389126/document
- See also: Mamadou Dia et al. A Novel Stochastic Transformer-based Approach for Post-Traumatic Stress Disorder Detection using Audio Recording of Clinical Interviews, CBMS, June 2023. — https://ieeexplore.ieee.org/document/10178722
- See also: J. Gratch et al. The Distress Analysis Interview Corpus of Human and Computer Interviews. — https://aclanthology.org/L14-1421/
- See also: X. Kong et al. Automatic Identification of Depression Using Facial Images with Deep Convolutional Neural Network. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9281460/
- See also: Mundt JC, Vogel AP, Feltner DE, Lenderking WR. Vocal acoustic biomarkers of depression severity and treatment response. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3409931/